CLINICAL TRIAL: NCT00446537
Title: Procedural Learning in Participants With ADHD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 240446
Record Dates: First submitted 2007-03-11; First posted 2007-03-13 (Estimated); Last update posted 2007-03-13 (Estimated); Status verified 2007-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Skill Acquisition and the Evolution of Long Term Procedural Memory in participants with ADHD: The Effect of Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Methylphenidate

SUMMARY:
Skill acquisition refers to the process of improvement of performance following practice experience. This process is the basis for generation of a long-lasting memory. Individuals with Attention Deficit Hyperactivity Disorder (ADHD) have been shown to be impaired on some performance aspects of previously learned skills, an impairment that is often ameliorated, at least temporarily, by psychostimulant medication (the standard therapy in ADHD). The proposed study aims to define the course of learning and of generation of long-term memory consolidation in individuals with ADHD, and to essay the effectiveness of psychostimulant medication on both the learning and retention of the skills.

DETAILED DESCRIPTION:
Skill Acquisition and the Evolution of Long Term Procedural Memory in participants with ADHD: The Effect of Methylphenidate

ELIGIBILITY:
Inclusion Criteria:

* Full scale IQ score of 85 or above

Ages: 12 Years to 50 Years | Sex: All
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Esther Adi-Japha, PhD, Principal Investigator — Bar-Ilan University, Israel; Ruth Shalev, MD, Study Chair — Shaare Zedek Medial Center
Locations (1):
- Neuropediatric Unit, Jerusalem, Israel